CLINICAL TRIAL: NCT05894759
Title: Psychodermatological Approaches of Psoriasis
Brief Title: The Impact of Different Relaxation Techniques on Psoriasis Patients With an Elevated Psychological Stress Level
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grigore T. Popa University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Bogdan-Marian Tarcau, Principal investigator, Grigore T. Popa University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 293/14.04.2023
Record Dates: First submitted 2023-05-17; First posted 2023-06-08 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Psoriasis; Stress, Psychological; Depression; Anxiety
MeSH Terms: conditions — Psoriasis; Stress, Psychological; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music therapy (Experimental): Patients will undergo music therapy, delivered online, for 1 month.
  Interventions: Behavioral: Psychological stress relief techniques
- Relaxing stories (Sham Comparator): Patients will listen to relaxing stories, online, for 1 month.
  Interventions: Behavioral: Psychological stress relief techniques
- Treatment as usual (No Intervention): Dermatological treatment as per national guidelines.

INTERVENTIONS:
Behavioral: Psychological stress relief techniques — Psychological stress relief techniques
  Arms: Music therapy; Relaxing stories

SUMMARY:
Two mind-relaxing techniques will be applied to psoriasis patients with an elevated psychological stress profile at baseline

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of psoriasis
* adequate psychological stress profile
* access to a personal computer/ laptop/ smartphone with internet connection
* agreement to the informed consent form

Exclusion Criteria:

* other dermatological conditions which impair the life quality
* psychological disorders under psychiatric treatment
* hearing impairment
* other on-going medical studies
* pregnancy
* aliteracy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Dermatological Life Quality Index | 6 months
  Dermatological Life Quality Index Score will be calculated at baseline, 1 month and 6 months.
  Dermatological Life Quality Index minimum score = 0 (no impairment of life quality) Dermatological Life Quality Index maximum score = 30 (maximum impairment of life quality)
Psychological stress | 6 months
  A visual analog scale will be used at baseline, 1 month and 6 months. Analog scale minimum value = 0 (no stress) Analog scale maximum value = 10 (maximum stress)
General Anxiety Disorder-7 | 6 months
  General Anxiety Disorder-7 questionnaire will be applied at baseline, 1 month and 6 months.
  General anxiety disorded-7 minimum score = 0 (no anxiety) General anxiety disorded-7 maximum score = 21 (maximum anxiety)
Patient Health Questionnaire-9 | 6 months
  Patient Health Questionnaire-9 will be applied at baseline, 1 month and 6 months.
  Patient Health Questionnaire-9 minimum score = 0 (no depression) Patient Health Questionnaire-9 maximum score = 27 (maximum depression)

SECONDARY OUTCOMES:
Psoriasis Area and Severity Index | 6 months
  Psoriasis Area and Severity Index score will be calculated will be applied at baseline, 1 month and 6 months.
  Psoriasis Area and Severity Index minimum score = 0 (no severity - no lesions) Psoriasis Area and Severity Index maximum score = 72 (maximum severity)
Self Administered Psoriasis Area and Severity Index | 6 months
  The self Administered Psoriasis Area and Severity Index score will be calculated by the patient at baseline, 1 month and 6 months.
  The self Administered Psoriasis Area and Severity Index minimum score = 0 (no severity - no lesions) The self Administered Psoriasis Area and Severity Index maximum score = 72 (maximum severity)
The Revised Illness Perception Questionnaire | 6 months
  The Revised Illness Perception Questionnaire will be applied at baseline, 1 month and 6 months.
  The Revised Illness Perception Questionnaire minimum score = 0 (best illness perception) The Revised Illness Perception Questionnaire maximum score = 80 (worst illness perception)
Dermatological treatment compliance | 6 months
  A visual analog scale will be applied at baseline, 1 month and 6 months. Analog scale minimum value = 0 (total lack of compliance) Analog scale maximum value = 10 (maximum compliance)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Gheuca Solovastru, Prof., Study Director — Grigore T. Popa University of Medicine and Pharmacy Iasi
Locations (1):
- Saint Spiridon Emergency Clinical County Hospital- Dermatology department, Iași, Romania

IPD SHARING:
Plan to Share IPD: No